CLINICAL TRIAL: NCT02310048
Title: A Randomised, Open-Label, Single-Dose, Parallel Group Study to Assess the Comparative Oral Bioavailability of Two Capsule Formulations of MT-1303 in Healthy Male Subjects
Brief Title: Comparative Oral Bioavailability Study of MT-1303
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-E09
Record Dates: First submitted 2014-11-14; First posted 2014-12-05 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

ARMS (2):
- MT-1303-FormA (Experimental): MT-1303, Capsule Formulation A
  Interventions: Drug: MT-1303-FormA
- MT-1303-FormB (Experimental): MT-1303, Capsule Formulation B
  Interventions: Drug: MT-1303-FormB

INTERVENTIONS:
Drug: MT-1303-FormA
  Arms: MT-1303-FormA
Drug: MT-1303-FormB
  Arms: MT-1303-FormB

SUMMARY:
The purpose of this study is to assess the comparative oral bioavailability of a Formulation B versus the Formulation A of MT-1303.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males aged 18 to 55 years at Screening.
* Healthy and free from clinically significant illness or disease as determined by medical history, physical examination, laboratory, and other tests at Screening and Day -1.
* A body weight of ≥60 kilograms (kg) and BMI ranging from 18 to 30 kg/m2 at Screening or Day -1.

Exclusion Criteria:

* Presence or history of severe adverse reaction or allergy to any medicinal product or relevant excipient that is of clinical significance.
* Participated in more than three clinical studies of a new chemical entity in the previous year or participated in a clinical study of any IMP within 12 weeks or five half-lives of the IMP before the administration of the IMP in this clinical study.
* Clinically relevant abnormal medical history, physical findings, or laboratory values at Screening or Day -1 that could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator.
* Previous medical history of tuberculosis or in the opinion of the Investigator a recurrent medical history of cold sores, pharyngitis, urinary tract infection, diarrhoea/dysentery, chest infections, or fungal infection.
* Subjects who have received any prescribed systemic or topical medication within 14 days prior to administration of the IMP(Day 1) unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety. Slow release medicinal formulations considered to still be active within 14 days prior to the first dose administration will also be excluded unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise safety.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve(AUC) . | up to 6 weeks

SECONDARY OUTCOMES:
Peak drug concentration (Cmax) of MT-1303 | up to 6 weeks
Time to reach peak concentration (Tmax) of MT-1303 | up to 6 weeks
Half-life(t1/2.) of MT-1303 | up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, Dr., Principal Investigator — Covance CRU Ltd.
Locations (1):
- Investigational site, Leeds, United Kingdom